CLINICAL TRIAL: NCT01413295
Title: Randomized Phase II Trial in Patients With Progressive Stage IV Colorectal Cancer to Two Lines of Chemotherapy, in Order to Compare the Best Supportive Treatment Versus Treatment With Dendritic Cells Plus the Best Supportive Treatment
Brief Title: Randomized Trial With Dendritic Cells in Patients With Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fundacion Clinic per a la Recerca Biomédica (Other)
Responsible Party: Principal Investigator, Ramon Vilella Puig, Senior consultant, Fundacion Clinic per a la Recerca Biomédica
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCBRVP; 2009-017247-33 (EudraCT Number); TRA-082 (Other Grant/Funding Number: Ministerio Ciencia e Innovación. SPAIN)
Record Dates: First submitted 2011-08-09; First posted 2011-08-10 (Estimated); Last update posted 2014-11-04 (Estimated); Status verified 2014-11

CONDITIONS: Colorectal Neoplasms
Keywords: Colorectal Neoplasms; Dendritic Cells
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dendritic Cells Vaccine (Experimental): Dendritic Cells Vaccine after 2 lines of chemotherapy
  Interventions: Drug: Dendritic Cell Vaccine
- Supportive treatment (Other): Supportive treatment after 2 lines of chemotherapy
  Interventions: Other: Supportive treatment

INTERVENTIONS:
Drug: Dendritic Cell Vaccine — Vaccination with autologous dendritic cells loaded with autologous tumor antigens
  Arms: Dendritic Cells Vaccine
Other: Supportive treatment — Supportive treatment after progression of the illness after 2 lines of chemotherapy
  Arms: Supportive treatment

SUMMARY:
The different alternatives used since 1996 to treat metastatic colorectal cancer (MCRC) have increased the mean survival of these patients. This outstanding advance is due to the extended indications for resection of hepatic metastases and to the use of new chemotherapeutic drugs (fluoropyrimidine, irinotecan and oxaliplatin) and monoclonal antibodies (bevacizumab, cetuximab and panitumumab). However, none of these treatments is curative and the majority of patients are overwhelmed by the illness. The first line of treatment for MCRC is FOLFOX and the second, irinotecan plus cetuximab for patients with wild type KRAS gene (60%) with a 30% responses, and bevacizumab plus irinotecan with a 5-10% of responses, in patients with mutated KRAS (40%). A treatment with autologous dendritic cells (DCs) pulsed with autologous tumour antigens is proposed as a third line of therapy. A randomized phase II trial would be performed, by selecting two groups of patients, one of them would be treated with the best supportive treatment and the other with DCs plus the best supportive treatment. The aim of the study would be to analyze the outcome after 4 months of treatment. In patients treated with DCs, IFN-γ spot forming cells and proliferative responses would be determined pre and post treatment in lymphocytes stimulated with autologous DCs pulsed with autologous tumour antigens. Pre and post treatment serum levels of IFN-γ, TNF-α, TGF-β e IL-12, would also be measured.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years.
* Capacity of understanding and signing the informed consent and to undergo the study procedures.
* Previously treated with 2 lines of chemotherapy.
* ECOG <= 2.
* Adequate renal, hepatic and bone marrow function
* Confirmed diagnosis of colorectal cancer with hepatic metastasis, suitable for biopsy.
* Availability of tumor tissue, for maturing dendritic cells
* RECIST.1 criteria

Exclusion Criteria:

* Clinically relevant diseases or infections (HBV, HCV, HIV).
* Pregnant or breast feeding women.
* Immunosuppressant treatment.
* Concurrent cancer, with the exceptions allowed by the principal investigator (PI).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2011-08; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival | 4 months

SECONDARY OUTCOMES:
Overall Survival | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Ramon Vilella, PhD, Principal Investigator — Fundació Clinic Recerca Biomédica
Locations (1):
- Hospital Clínic Barcelona, Barcelona, Barcelona, Spain